CLINICAL TRIAL: NCT04396366
Title: A Randomized, Subject- and Investigator-blinded, Placebo-controlled, Parallel Group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of QBW251 in Patients With Bronchiectasis
Brief Title: Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of QBW251 in Subjects With Bronchiectasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic business decision
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQBW251C12201
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; QBW251; colony forming units
MeSH Terms: conditions — Bronchiectasis | interventions — icenticaftor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QBW251 300 mg b.i.d (Experimental): Participants received QBW251 300 mg orally, twice daily (b.i.d.), for 12 weeks.
  Interventions: Drug: QBW251
- Placebo (Placebo Comparator): Participants received matching placebo, b.i.d., for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QBW251 — QBW251, 300 mg, oral use, one capsule, twice daily.
  Arms: QBW251 300 mg b.i.d
Drug: Placebo — Matching placebo, 300 mg, oral use, one capsule, twice daily.
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether potentiating the cystic fibrosis transmembrane conductance regulator (CFTR) with QBW251 in patients with bronchiectasis will demonstrate clinical safety and efficacy related to improved mucociliary clearance with reduced bacterial colonization as potential drivers of airway obstruction, reduced airway inflammation, exacerbations and mucus load, improved lung function, clinical symptoms and quality of life to support further development in bronchiectasis.

DETAILED DESCRIPTION:
This was a randomized, participant- and investigator-blinded, placebo-controlled, parallel-group study investigating the preliminary efficacy and safety of QBW251 administered orally for 12 weeks in participants with bronchiectasis. Approximately 72 subjects were planned to be randomized in a 1:1 ratio to receive either QBW251 or placebo in order to achieve 60 subjects to complete the treatment period based on the assumption of a 16% drop-out rate. However, the study was prematurely terminated due to a Novartis strategic decision. As a result, only 42 participants were randomized to either the QBW251 300 mg b.i.d group or the placebo group.

The study consisted of the screening, baseline/Day 1, treatment period, and end of study assessments (EOS) visit followed by an additional post-treatment safety follow up via phone call. The total duration for each patient in the study was up to approximately 19 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years at screening.
* Proven diagnosis of bronchiectasis by chest CT at screening as determined by investigator.
* Evidence of sputum bacterial load of ≥106 CFU/mL with at least one potentially pathogenic microorganism (H. Influenzae, M catarrhalis, S aureus, S pneumoniae, Enterobacteriaceae, P aeruginosa, Stenotrophomonous maltophilia, or any potential pathogenic non-fermenting Gram-negative bacteria measured by dilution/outgrowth).
* Documented history of at least one bronchiectasis exacerbation between January 2019 and study screening.
* Patients with bronchial hypersecretion, defined as productive cough that occurred on most days (defined as >50% days) for at least three consecutive months within 12 months prior to screening, as assessed by documentation of patient recollection (anamnesis) or documented in patients' record.
* Patients were allowed to stay on fixed or free combinations of LABA/LAMA or LABA/ICS or LABA/LAMA/ICS as maintenance therapy if they were treated with them at a stable dose for the last 3 months prior to screening. Patients were also allowed to stay on macrolides as maintenance therapy if they were treated with them at a stable dose, 3 months before screening. Patients were allowed to use mucolytics or hyperosmolar agents if they were treated with them before study start.
* If prescribed, patients were included in the study with unchanged chest physiotherapy for at least 4 weeks prior to screening.
* Clinically stable pulmonary status in the opinion of the investigator and unlikely to require any change in the standard regimen of care during the course of the study.

Exclusion Criteria:

* Patients with a history of long-QT syndrome or the QTcF interval at screening and baseline was prolonged (QTcF > 450 ms in males, > 460 ms in females).
* Patients with a history or current treatment for hepatic disease including but not limited to acute or chronic hepatitis, cirrhosis or hepatic failure. A history of resolved Hepatitis A was not exclusionary. Patients with a prothrombin time international normalized ratio (PT/INR) of more than 1.5 × ULN at screening. Patients excluded for the PT/INR of more than 1.5 x ULN could be re-screened when the values returned to normal.
* History of lung transplant or malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there was evidence of local recurrence or metastases. Patients with segmentectomy for other reasons than cancer were allowed to be included in the study. Patients with a history of cancer and 5 years or more disease free survival time might be included in the study by agreement with Novartis Medical Monitor on a case-by-case basis.
* Patients requiring long-term oxygen therapy for chronic hypoxemia. This was typically patients requiring oxygen therapy >12 h per day delivered by home oxygen cylinder or concentrator. Note: Nocturnal oxygen therapy for transient oxygen desaturations during sleep was allowed.
* Patients with bronchiectasis who had a pulmonary exacerbation with a deterioration in three or more of the following key symptoms for at least 48 h:

  * cough;
  * sputum volume and/or consistency;
  * sputum purulence;
  * breathlessness and/or exercise tolerance;
  * fatigue and/or malaise;
  * hemoptysis And A clinician determined that a change in bronchiectasis treatment was required (e.g., requiring systemic glucocorticosteroid treatment and/or systemic or inhaled antibiotics) within 4 weeks prior to screening.

In the event of an exacerbation occurring 4 weeks before screening, or between the screening and baseline (please see definition above), the participant was not to be enrolled. The participant might be rescreened once, 4 weeks after the resolution of exacerbation.

* Participants with bronchiectasis requiring therapy that might interfere with the assessment of QBW251 efficiency or who were unlikely to respond to QBW251 as follows:
* Participants with suspected active pulmonary tuberculosis or currently being treated for active pulmonary tuberculosis were not allowed. Note: Participants with a history of pulmonary tuberculosis could be enrolled if they met the following requirements: history of appropriate drug treatment followed by negative imaging results within 12 months prior to baseline visit suggesting low probability of recurrent active tuberculosis
* Patients with active allergic bronchopulmonary aspergillosis and asthma as primary diagnosis.
* Patients with cystic fibrosis
* Current or ex-smokers with severe emphysema.
* Participants with another concomitant pulmonary disease according to the definition of the International ERS/ATS guidelines, including but not limited to idiopathic pulmonary fibrosis (IPF), sarcoidosis or other granulomatous or infectious process. Concomitant COPD and asthma with characteristics of airway hyperresponsiveness as well as COPD-Asthma overlap syndrome were allowed as long as it was not the main, primary diagnosis in the opinion of the investigator. Primary ciliary dyskinesia (PCD) was allowed.
* Participants currently receiving treatment for nontuberculous mycobacterial (NTM) pulmonary disease. If performed, patients with one or more positive cultures in the last 12 months for M. avium complex, M. abscessus complex, M. kansasii, M. malmoense, M. xenopi, M. simiae or M. chelonae, unless all subsequent NTM cultures (at least two) were negative and in the opinion of the investigator the patient did not met ATS criteria for NTM-pulmonary disease.
* Patients receiving any medication that might influence the response to treatment within 4 weeks prior to screening including systemic or inhaled steroids (ICS alone), or other systemic immunomodulators, recombinant human DNAse, any systemic or inhaled antibiotics.
* Patients with a body mass index (BMI) of more than 40 kg/m^2

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- China (2):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shanghai
- Germany (3):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mainz
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
- United Kingdom (6):
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2456

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All inclusion and exclusion criteria were checked at screening.
Period: Overall Study
Arm/Group | QBW251 300 mg b.i.d | Placebo
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QBW251 300 mg b.i.d | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (15.80) | 56.2 (12.96) | 54.5 (14.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 10 | 11 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 11 | 10 | 21
  White | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Bacterial Load Colony-forming Units of Potentially Pathogenic Microorganisms in Sputum at Week 12
Description: This measure reflects the amount of bacteria present in a patient's lungs.
Time Frame: Baseline, 12 weeks
Population: The Pharmacodynamics (PD) Analysis Set included all participants with available PD data at both baseline and at least one post-baseline assessment that were not affected by any protocol deviations. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 13 | 19
CFU/mL | -0.192 (1.4621) | 0.340 (1.6476)

2. Secondary Outcome: Number of Participants With Absence of Any Colony-forming Units of Potentially Pathogenic Bacteria Sputum
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 21 | 21
Participants | 0 | 0

3. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B) (Respiratory Symptoms Domain)
Description: The Quality of Life Questionnaire for Bronchiectasis (QOL-B) is a disease-specific questionnaire developed for non-cystic fibrosis bronchiectasis. It covers 8 dimensions: physical functioning, role functioning, emotional functioning, social functioning, vitality, treatment burden, health perceptions, and respiratory symptoms. Each dimension is scored separately on a scale of 0 to 100, and higher scores represent better outcomes. Only the respiratory symptoms domain score is reported for this outcome measure.
Time Frame: Baseline, Days 28, 56, 84
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 13 | 20
score on a scale
  Day 28 n=12,19: number analyzed (Participants) | 12 | 19
  Day 28 n=12,19 | 5.247 (10.9936) | 7.212 (9.5209)
  Day 56 n=12,20: number analyzed (Participants) | 12 | 20
  Day 56 n=12,20 | 1.852 (5.8026) | 1.852 (11.7429)
  Day 84 n=13,20 | 2.849 (9.4612) | 3.519 (11.9848)

4. Secondary Outcome: Change From Baseline in Fibrinogen Plasma Concentration
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 19 | 19
g/L | -0.193 (0.6278) | -0.127 (0.4828)

5. Secondary Outcome: Change From Baseline in Daily Rescue Medication Use (Salbutamol/Albuterol)
Description: The total number of puffs of rescue medication was divided by the total number of (full or half) days with non-missing rescue data to derive the mean daily number of puffs of rescue medication taken for the patient for the given visit interval.
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: number of puffs
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 20
number of puffs | -0.37 (1.069) | 0.14 (0.895)

6. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Exploratory Volume in the First Second (FEV1)
Description: FEV1 is the amount of air that can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Baseline, Days 28, 56, 84
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 20 | 20
liters
  Day 28 n=20,20 | -0.002 (0.1113) | 0.012 (0.1541)
  Day 56 n=18,18: number analyzed (Participants) | 18 | 18
  Day 56 n=18,18 | 0.031 (0.1086) | 0.007 (0.1137)
  Day 84 n=17,19: number analyzed (Participants) | 17 | 19
  Day 84 n=17,19 | 0.045 (0.1650) | 0.022 (0.1260)

7. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Days 28, 56, 84
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 20 | 20
liters
  Day 28 n=20,20 | -0.068 (0.1834) | -0.017 (0.1685)
  Day 56 n=18,18: number analyzed (Participants) | 18 | 18
  Day 56 n=18,18 | -0.019 (0.1943) | -0.049 (0.1358)
  Day 84 n=17,19: number analyzed (Participants) | 17 | 19
  Day 84 n=17,19 | -0.019 (0.1779) | 0.034 (0.2156)

8. Secondary Outcome: Change From Baseline in Bronchus Region Pi10
Description: Pi10 is the square root of the wall area for an idealized airway with a luminal perimeter of 10 mm. Pi10 is the most commonly used measure of wall thickening and represents a regional estimate of the small airways across the whole lung or a particular lobe. Measured by high resolution computed tomography (HRCT).
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 21 | 21
mm
  Lung, Left, Inferior Lobe, Posterior Basal Segment n=21,21 | -0.072 (0.3592) | -0.029 (1456)
  Lung, Left, Superior Lobe, Apical Segment n=16,18: number analyzed (Participants) | 16 | 18
  Lung, Left, Superior Lobe, Apical Segment n=16,18 | -0.063 (0.4140) | 0.029 (0.1600)
  Lung, Right, Inferior Lobe, Posterior Basal Segment n=14,18: number analyzed (Participants) | 14 | 18
  Lung, Right, Inferior Lobe, Posterior Basal Segment n=14,18 | 0.001 (0.1999) | -0.015 (0.1071)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19: number analyzed (Participants) | 16 | 19
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | 0.074 (0.1867) | 0.039 (0.1471)
  Lung, Right, Superior Lobe, Apical Segment n=15,19: number analyzed (Participants) | 15 | 19
  Lung, Right, Superior Lobe, Apical Segment n=15,19 | -0.037 (0.1990) | -0.026 (0.0991)

9. Secondary Outcome: Change From Baseline in Region Percent Below or Equal to -856 Hounsfield Units (HU)
Description: The region percent below or equal to -856 HU represents air trapping, which was evaluated by HRCT in the whole lung and in the regions (thirds, lobes).
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: percent of region
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 15 | 17
percent of region
  Lung n=15,17 | -0.284 (9.2755) | -1.074 (8.7794)
  Lung, Left n=15,17 | -1.659 (8.5613) | -1.095 (7.2200)
  Lung, Left Lower Lobe n=15,17 | -3.582 (8.4976) | -2.975 (7.8007)
  Lung, Left Upper Lobe n=15,17 | 0.002 (10.3698) | 1.946 (10.7307)
  Lung, Right n=15,17 | 1.410 (10.8421) | -1.552 (10.1631)
  Lung, Right Lower Lobe n=15,17 | 0.303 (7.9933) | -2.193 (10.7784)
  Lung, Right Middle Lobe n=15,17 | 2.877 (10.3635) | 0.502 (9.3885)
  Lung, Right Upper Lobe n=15,17 | 1.513 (13.1404) | -2.105 (11.4788)
  Thirds, Left Lower n=15,17 | -2.726 (9.4063) | -1.109 (4.8754)
  Thirds, Left Middle n=15,17 | -2.319 (8.3145) | -0.892 (8.0664)
  Thirds, Left Upper n=15,17 | 0.940 (10.8083) | -1.056 (9.7966)
  Thirds, Right Lower n=15,17 | 0.394 (9.2444) | -2.214 (9.6626)
  Thirds, Right Middle n=15,17 | 1.563 (11.7119) | -0.804 (10.4909)
  Thirds, Right Upper n=15,17 | 1.905 (12.7615) | -2.052 (11.7677)

10. Secondary Outcome: Change From Baseline in Region Air Volume
Description: Measured by HRCT
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
liters
  Lung n=16,19 | 7.588 (362.231) | -4.667 (323.292)
  Lung, Left n=16,19 | 6.719 (188.304) | -7.304 (144.047)
  Lung, Left Lower Lobe n=15,19: number analyzed (Participants) | 15 | 19
  Lung, Left Lower Lobe n=15,19 | 22.142 (125.643) | -14.848 (84.4328)
  Lung, Left Upper Lobe n=16,19 | -14.039 (82.9500) | 7.545 (69.1768)
  Lung, Right n=16,19 | 0.869 (179.912) | 2.637 (190.892)
  Lung, Right Lower Lobe n=16,19 | 9.886 (95.0629) | -5.435 (105.079)
  Lung, Right Middle Lobe n=16,19 | -3.233 (20.4193) | 1.242 (13.5834)
  Lung, Right Upper Lobe n=16,19 | -5.784 (78.3195) | 6.830 (81.4095)
  Thirds, Left Lower n=16,19 | -3.409 (82.0621) | -5.155 (50.2945)
  Thirds, Left Middle n=16,19 | -1.319 (76.6437) | -1.992 (63.8795)
  Thirds, Left Upper n=16,19 | 11.444 (73.0426) | -0.432 (41.7288)
  Thirds, Right Lower n=16,19 | -20.490 (122.493) | -7.548 (76.9902)
  Thirds, Right Middle n=16,19 | 8.762 (98.3416) | 2.994 (93.2434)
  Thirds, Right Upper n=16,19 | 12.574 (84.6939) | 5.327 (60.5143)

11. Secondary Outcome: Change From Baseline in Segment Average Inner Area
Description: Measured by HRCT
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
mm^2
  Lower Lobe Bronchus, Left n=15,17: number analyzed (Participants) | 15 | 17
  Lower Lobe Bronchus, Left n=15,17 | 2.009 (10.4977) | -1.376 (6.5410)
  Lung, Left Upper Lobe n=15,18: number analyzed (Participants) | 15 | 18
  Lung, Left Upper Lobe n=15,18 | 1.106 (11.1387) | 1.506 (7.5668)
  Lung, Right Lower Lobe n=16,19 | -0.677 (7.9904) | -2.119 (6.7263)
  Lung, Right Upper Lobe n=16,19 | 0.667 (4.9950) | -2.653 (14.9922)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | 0.138 (4.8198) | -0.379 (2.8929)
  Lung, Right, Middle Lobe, Medial Segment n=16,19 | -0.502 (5.2215) | 1.828 (5.5992)

12. Secondary Outcome: Change From Baseline in Segment Average Major Inner Diameter
Description: Measured by HRCT
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
mm
  Lower Lobe Bronchus, Left n=15,17: number analyzed (Participants) | 15 | 17
  Lower Lobe Bronchus, Left n=15,17 | 0.364 (1.0234) | -0.128 (0.5242)
  Lung, Left Upper Lobe n=15,18: number analyzed (Participants) | 15 | 18
  Lung, Left Upper Lobe n=15,18 | -0.095 (0.7972) | -0.116 (0.7192)
  Lung, Right Lower Lobe n=16,19 | -0.040 (0.7883) | -0.207 (0.7876)
  Lung, Right Upper Lobe n=16,19 | 0.081 (0.7149) | -0.525 (1.9690)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | 0.075 (0.9001) | -0.066 (0.5419)
  Lung, Right, Middle Lobe, Medial Segment n=16,19 | 0.046 (0.8759) | 0.336 (1.2354)

13. Secondary Outcome: Change From Baseline in Segment Average Minor Inner Diameter
Description: Measured by HRCT
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
mm
  Lower Lobe Bronchus, Left n=15,17: number analyzed (Participants) | 15 | 17
  Lower Lobe Bronchus, Left n=15,17 | 0.080 (0.8100) | -0.204 (0.7995)
  Lung, Left Upper Lobe n=15,18: number analyzed (Participants) | 15 | 18
  Lung, Left Upper Lobe n=15,18 | 0.160 (0.7449) | 0.120 (0.5935)
  Lung, Right Lower Lobe n=16,19 | -0.011 (0.6186) | -0.220 (0.6556)
  Lung, Right Upper Lobe n=16,19 | 0.034 (0.4546) | 0.127 (0.5699)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | -0.037 (0.5225) | -0.058 (0.4702)
  Lung, Right, Middle Lobe, Medial Segment n=16,19 | -0.309 (0.7621) | 0.065 (0.5016)

14. Secondary Outcome: Change From Baseline in Segment Average Outer Area
Description: Measured by HRCT
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
mm^2
  Lower Lobe Bronchus, Left n=15,17: number analyzed (Participants) | 15 | 17
  Lower Lobe Bronchus, Left n=15,17 | 3.805 (15.3509) | -3.575 (9.6603)
  Lung, Left Upper Lobe n=15,18: number analyzed (Participants) | 15 | 18
  Lung, Left Upper Lobe n=15,18 | 2.527 (25.2783) | 6.387 (15.1487)
  Lung, Right Lower Lobe n=16,19 | -0.887 (13.2296) | -2.439 (10.4313)
  Lung, Right Upper Lobe n=16,19 | 3.054 (11.6503) | -6.171 (35.7465)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | 0.011 (8.9779) | -0.574 (6.6601)
  Lung, Right, Middle Lobe, Medial Segment n=16,19 | -1.929 (12.3065) | 3.655 (9.0492)

15. Secondary Outcome: Change From Baseline in Segment Average Wall Area Fraction
Description: Wall area fraction or ratio was calculated by dividing the wall area of the corresponding segment to the total airway area. Measured by HRCT.
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
ratio
  Lower Lobe Bronchus, Left n=15,17: number analyzed (Participants) | 15 | 17
  Lower Lobe Bronchus, Left n=15,17 | -0.009 (0.0515) | -0.002 (0.0310)
  Lung, Left Upper Lobe n=15,18: number analyzed (Participants) | 15 | 18
  Lung, Left Upper Lobe n=15,18 | 0.002 (0.0553) | 0.013 (0.0436)
  Lung, Right Lower Lobe n=16,19 | 0.001 (0.0377) | 0.011 (0.0277)
  Lung, Right Upper Lobe n=16,19 | 0.007 (0.0392) | 0.001 (0.0347)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | -0.002 (0.0414) | 0.006 (0.0262)
  Lung, Right, Middle Lobe, Medial Segment n=16,19 | 0.007 (0.0281) | 0.002 (0.0347)

16. Secondary Outcome: Change From Baseline in Segment Average Wall Thickness
Description: Measured by HRCT
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
mm
  Lower Lobe Bronchus, Left n=15,17: number analyzed (Participants) | 15 | 17
  Lower Lobe Bronchus, Left n=15,17 | 0.001 (0.1680) | -0.042 (0.0987)
  Lung, Left Upper Lobe n=15,18: number analyzed (Participants) | 15 | 18
  Lung, Left Upper Lobe n=15,18 | 0.014 (0.3422) | 0.081 (0.2417)
  Lung, Right Lower Lobe n=16,19 | 0.001 (0.1691) | 0.021 (0.0900)
  Lung, Right Upper Lobe n=16,19 | 0.054 (0.2231) | -0.030 (0.2941)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | -0.014 (0.0828) | -0.004 (0.0968)
  Lung, Right, Middle Lobe, Medial Segment n=16,19 | -0.040 (0.1606) | 0.057 (0.0766)

17. Secondary Outcome: Change From Baseline in Segment Wall Area Percent
Description: Measured by HRCT
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
percent
  Lower Lobe Bronchus, Left n=15,17: number analyzed (Participants) | 15 | 17
  Lower Lobe Bronchus, Left n=15,17 | -0.009 (0.0515) | -0.002 (0.0305)
  Lung, Left Upper Lobe n=15,18: number analyzed (Participants) | 15 | 18
  Lung, Left Upper Lobe n=15,18 | 0.002 (0.0553) | 0.013 (0.0437)
  Lung, Right Lower Lobe n=16,19 | 0.001 (0.0376) | 0.011 (0.0276)
  Lung, Right Upper Lobe n=16,19 | 0.007 (0.0394) | 0.002 (0.0337)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | -0.003 (0.0411) | 0.006 (0.0261)
  Lung, Right, Middle Lobe, Medial Segment n=16,19 | 0.007 (0.0282) | 0.002 (0.0347)

18. Secondary Outcome: Change From Baseline in Segment Wall Area
Description: Measured by HRCT
Time Frame: Baseline, 12 weeks
Population: PD Analysis Set. Results are reported for participants with available data.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | QBW251 300 mg b.i.d | Placebo
Number analyzed (Participants) | 16 | 19
mm^2
  Lower Lobe Bronchus, Left n=15,17: number analyzed (Participants) | 15 | 17
  Lower Lobe Bronchus, Left n=15,17 | 1.796 (6.6301) | -2.199 (4.3938)
  Lung, Left Upper Lobe n=15,18: number analyzed (Participants) | 15 | 18
  Lung, Left Upper Lobe n=15,18 | 1.421 (18.5698) | 4.881 (12.4380)
  Lung, Right Lower Lobe n=16,19 | -0.209 (6.9730) | -0.320 (4.5446)
  Lung, Right Upper Lobe n=16,19 | 2.388 (9.7223) | -3.518 (21.8864)
  Lung, Right, Middle Lobe, Lateral Segment n=16,19 | -0.127 (4.6312) | -0.194 (4.0452)
  Lung, Right, Middle Lobe, Medial Segment n=16,19 | -1.427 (7.3051) | 1.827 (3.8885)

19. Secondary Outcome: Cmax of QBW251
Description: Maximum (peak) plasma concentration of QBW251
Time Frame: 1h, 2h, 3h, 4h, 6h and 8h post-dose on Days 1 and 28, and 3h post-dose on Day 56 and Day 84
Population: The pharmacokinetic (PK) analysis set included all participants with at least one available valid PK concentration measurement, who received any dose of QBW251 and had no protocol deviations that affected PK data. PK parameters were only analyzed in the QBW251 arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 300 mg b.i.d
Number analyzed (Participants) | 19
ng/mL
  Day 1 n=19 | 1120 (913)
  Day 28 n=19 | 1520 (951)
  Day 56 n=19 | 1190 (578)
  Day 84 n=18: number analyzed (Participants) | 18
  Day 84 n=18 | 1460 (947)

20. Secondary Outcome: Ctrough of QBW251
Description: Trough (pre-dose) plasma concentration of QBW251
Time Frame: Pre-dose Day 1, Day 28, Day 56, Day 84
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 300 mg b.i.d
Number analyzed (Participants) | 21
ng/mL
  Day 1 n=21 | 0.00 (0.00)
  Day 28 n=20: number analyzed (Participants) | 20
  Day 28 n=20 | 489 (371)
  Day 56 n=19: number analyzed (Participants) | 19
  Day 56 n=19 | 483 (395)
  Day 84 n=18: number analyzed (Participants) | 18
  Day 84 n=18 | 498 (416)

21. Secondary Outcome: Cmax of QBW251 for a Serial PK Set
Time Frame: Pre-dose, 1h, 2h, 3h, 4h, 6h and 8h post-dose on Day 1 and Day 28
Population: The pharmacokinetic (PK) analysis set included all participants with at least one available valid PK concentration measurement, who received any dose of QBW251 and had no protocol deviations that affected PK data. Results data were collected for a subset of participants at selected sites. PK parameters were only analyzed in the QBW251 arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 300 mg b.i.d
Number analyzed (Participants) | 3
ng/mL
  Day 1 | 2470 (787)
  Day 28 | 3000 (1390)

22. Secondary Outcome: Ctrough of QBW251 for a Serial PK Set
Time Frame: Pre-dose, 1h, 2h, 3h, 4h, 6h and 8h post-dose on Day 1 and Day 28
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 300 mg b.i.d
Number analyzed (Participants) | 3
ng/mL
  Day 1 | 0.00 (0.00)
  Day 28 | 603 (142)

23. Secondary Outcome: AUClast of QBW251 for a Serial PK Set
Description: Area under the concentration-time curve up to the last measurable concentration of QBW251 (AUClast)
Time Frame: Pre-dose, 1h, 2h, 3h, 4h, 6h and 8h post-dose on Day 1 and Day 28
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | QBW251 300 mg b.i.d
Number analyzed (Participants) | 3
h*ng/mL
  Day 1 | 6100 (2340)
  Day 28 | 10300 (3100)

24. Secondary Outcome: Tmax of QBW251 for a Serial PK Set
Description: Time to reach maximum (peak) plasma concentration after single-dose administration
Time Frame: Pre-dose, 1h, 2h, 3h, 4h, 6h and 8h post-dose on Day 1 and Day 28
Population: as for outcome 21
Measure: Median (Full Range); unit: hours
Arm/Group | QBW251 300 mg b.i.d
Number analyzed (Participants) | 3
hours
  Day 1 | 1.00 [1.00 to 4.00]
  Day 28 | 2.00 [1.00 to 3.08]

25. Secondary Outcome: AUC0-12h of QBW251 for a Serial PK Set
Description: Twelve-hour AUC
Time Frame: Pre-dose, 1h, 2h, 3h, 4h, 6h and 8h post-dose on Day 1 and Day 28
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | QBW251 300 mg b.i.d
Number analyzed (Participants) | 2
h*ng/mL
  Day 1 n=2 | 5260 (1780)
  Day 28 n=1: number analyzed (Participants) | 1
  Day 28 n=1 | 15400 (NA) — Not calculable due to the single participant data point.

26. Secondary Outcome: Tlast of QBW251 for a Serial PK Set
Description: Tlast is the last measurable concentration sampling time.
Time Frame: Pre-dose, 1h, 2h, 3h, 4h, 6h and 8h post-dose on Day 1 and Day 28
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | QBW251 300 mg b.i.d
Number analyzed (Participants) | 3
hours
  Day 1 | 7.99 (0.00962)
  Day 28 | 8.00 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post-treatment, up to a maximum duration of 114 days.
Groups:
- Total: Total
Arm/Group | QBW251 300 mg b.i.d | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/42
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/21 | 2/42
Other Adverse Events (participants affected / at risk) | 14/21 | 13/21 | 27/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QBW251 300 mg b.i.d (N=21) | Placebo (N=21) | Total (N=42)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QBW251 300 mg b.i.d (N=21) | Placebo (N=21) | Total (N=42)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 2
Fatigue (General disorders) | 3 | 5 | 8
Peripheral swelling (General disorders) | 0 | 2 | 2
Pyrexia (General disorders) | 3 | 1 | 4
COVID-19 (Infections and infestations) | 3 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4
Dizziness (Nervous system disorders) | 3 | 0 | 3
Headache (Nervous system disorders) | 2 | 2 | 4
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT04396366/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT04396366/SAP_001.pdf